CLINICAL TRIAL: NCT00769015
Title: Low Vision Depression Prevention Trial for Age Related Macular Degeneration
Acronym: VITAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1U01EY018819 (NIH)
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Age-related Macular Degeneration; Depression
Keywords: age-related macular degeneration; depression; vision loss
MeSH Terms: conditions — Macular Degeneration; Depression; Vision Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BA-LVR (Experimental): In BA-LVR, a low vision occupational therapist (OT) will deliver Behavior Activation (BA), a psychological treatment to prevent depression. This will be administered in the context of the standard of low vision care for OTs as defined by the American Occupational Therapy Association (AOTA). The OTs will collaborate with low vision optometrists, who will deliver the standard of low vision care as defined by the American Optometric Association. The optometrists will evaluate remaining vision and magnification needs, prescribe optical devices, and provide the OTs with initial care plans. The OTs will subsequently meet with subjects in their homes 6 times over 12 weeks to enhance device use, home modifications, and compensatory strategies.
  Interventions: Behavioral: BA-LVR
- ST-LVR (Placebo Comparator): Subjects randomized to ST-LVR will receive clinic-based low vision optometry, in addition to 6 in-home Supportive Therapy (ST) sessions. ST is a placebo condition that controls for the attention that subjects in the active treatment arm will receive.
  Interventions: Behavioral: ST-LVR

INTERVENTIONS:
Behavioral: BA-LVR — Low vision clinic-based optometry plus 6 in-home occupational therapy visits
  Arms: BA-LVR
Behavioral: ST-LVR — Clinic-based low vision optometry plus 6 in-home sessions of Supportive Therapy
  Arms: ST-LVR

SUMMARY:
This randomized, controlled clinical trial, the Low Vision Depression Prevention TriAL (VITAL), will test the efficacy of collaborative low vision rehabilitation (LVR) to prevent depressive disorders in Age-Related Macular Degeneration (AMD). In this innovative intervention, a low vision occupational therapist collaborates with a low vision optometrist to develop and implement a care plan based on a subject's vision status, rehabilitation potential, and personal rehabilitation goals. An independent rater masked to treatment assignment will assess depressive disorders meeting DSM-IV criteria (primary outcome) and targeted vision function and vision-related quality of life (secondary outcomes) at baseline and then at 4 months to evaluate short-term effects (main trial end point) and at 12 months to evaluate long-term effects.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of blindness in older persons in the U.S. and affects more than 10 million people. One third of patients with AMD become clinically depressed when they lose the ability to pursue valued activities. Because their depression is disabling and unlikely to be treated, preventing depression in AMD is a public health imperative as the population ages.

We will recruit 200 subjects who have bilateral AMD and subthreshold depressive symptoms. Their bilateral vision loss and subthreshold depressive symptoms increase their risk to develop more severe depressive disorders and functional decline. We will randomize eligible subjects to collaborative Low Vision Rehabilitation (LVR) (optometrist and home-based OT) or enhanced LVR (optometrist and home-based Supportive Therapy). In this study, usual care LVR is enhanced with Supportive Therapy (ST), which is a standardized placebo psychological treatment that controls for attention.

Many older persons with AMD understandably become depressed when their vision loss prevents them from pursuing valued goals. This necessitates a disease management strategy that combines treatment for vision loss and depression. Because depression in AMD is rarely treated, preventing depression is more sensible than waiting to treat it after diagnosis or failing to treat it at all. As the population ages and more people are affected with AMD, finding ways to prevent depression and improve daily functioning has great public health importance. For these reasons, the VITAL Trial has high clinical significance to patients with AMD, and wider public health significance as our society confronts the challenge of caring for the growing population of older adults with chronic disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 65 years old
* Bilateral AMD
* Subthreshold depressive symptoms
* At least 1 vision goal that is important yet difficult to carry out

Exclusion Criteria:

* Uncontrolled glaucoma, diabetic retinopathy, corneal dystrophy, or cataracts for which surgery within 6 months is likely will be exclusionary conditions
* Current diagnosis of depression
* Cognitive impairment
* Life-threatening illness or any other health conditions that interferes with study activities.
* Patients who have received low vision rehabilitation or home-based OT in the preceding 12 months will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 188 (Actual)
Dates: Start 2009-06; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Rovner BW, Casten RJ, Hegel MT, Massof RW, Leiby BE, Ho AC, Tasman WS. Low vision depression prevention trial in age-related macular degeneration: a randomized clinical trial. Ophthalmology. 2014 Nov;121(11):2204-11. doi: 10.1016/j.ophtha.2014.05.002. Epub 2014 Jul 9. PMID 25016366
- [Derived] Deemer AD, Massof RW, Rovner BW, Casten RJ, Piersol CV. Functional Outcomes of the Low Vision Depression Prevention Trial in Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2017 Mar 1;58(3):1514-1520. doi: 10.1167/iovs.16-20001. PMID 28273318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from July 2009 through Feb 2013 from a large, private retina practice.
Period: Overall Study
Arm/Group | BA-LVR | ST-LVR
Started | 96 | 92
Completed | 87 | 76
Not Completed | 9 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BA-LVR | ST-LVR | Total
Number analyzed (Participants) | 96 | 92 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.2 (6.6) | 82.7 (6.9) | 84.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 62 | 132
  Male | 26 | 30 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 94 | 90 | 184
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 95 | 92 | 187
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: The primary outcome was a DSM-IV diagnosis of major or minor depression based on the Patient Health Questionnaire-9 (PHQ-9).13 The PHQ-9 includes the 9 criteria that define DSM-IV diagnoses of depression and is valid in low-vision patients. A scoring algorithm determines whether the profile of symptoms meets categorical diagnoses of depression. The model is adjusted for treatment group, vision stratum (20/70 to 20/100 vs. < 20/100), baseline better eye scotoma size, baseline depression scores [Patient Health Questionnaire (PHQ-9)], Medical Outcome Study score (MOS-6), which is a global index of self-rated physical and mental health, and baseline neuroticism scores.
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | BA-LVR | ST-LVR
Number analyzed (Participants) | 87 | 76
participants
  Total Sample | 11 | 18
  Worse Vision Group (< 20/100) | 5 | 11
  Better Vision Group (20/70 to 20/100) | 6 | 7
Statistical Analysis 1: Comparison: BA-LVR vs ST-LVR; Test type: Superiority or Other; p = .067, Mantel Haenszel — Mantel-Haenszel chi-square test. The p-value refers to the overall test of between group differences in rates of depression; Risk Ratio (RR) = .54, 95% CI 2-sided [.27 to 1.06]

2. Secondary Outcome: Vision Function: Distance Activities
Description: Distance vision function was assessed using the near activities subscale of the National Eye Institute Vision Function Questionaire-25 (NEI-VFQ). This subscale measures self-reported difficulty in completing activities that require distance function. The subscale is scored from 0 to 100 with higher scores indicating better function. Changes in least squares mean (95% CI) from month 0 to month 4 are reported.
Time Frame: 4 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BA-LVR | ST-LVR
Number analyzed (Participants) | 87 | 76
units on a scale | 0.31 [-3.25 to 3.87] | 1.12 [-2.54 to 4.78]
Statistical Analysis 1: Comparison: BA-LVR vs ST-LVR; Test type: Superiority or Other; p = .75, Linear Mixed effects model; Mean Difference (Net) = -.81, 95% CI 2-sided [-5.92 to 4.30]

3. Secondary Outcome: Quality of Life: Dependency
Description: Self-reported depencency was assessed using the Dependency subscale from the National Eye Institute Vision Function Questionaire-25 (NEI-VFQ). Scores range from 0 to 100, with higher scores indicating less dependency. Changes in least square means from baseline to 4 months are presented.
Time Frame: 4 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BA-LVR | ST-LVR
Number analyzed (Participants) | 87 | 76
units on a scale | 2.07 [-4.03 to 8.18] | 5.54 [-0.73 to 11.81]
Statistical Analysis 1: Comparison: BA-LVR vs ST-LVR; Test type: Superiority or Other; p = .68, Mixed Models Analysis; Change in least squares mean = 3.47, 95% CI 2-sided [-12.22 to 5.29]

4. Secondary Outcome: Vision Function: Near Activities
Description: Near vision function was assessed using the near activities subscale of the National Eye Institute Vision Function Questionaire-25 (NEI-VFQ). This subscale measures self-reported difficulty in completing activities that require near function. The subscale is scored from 0 to 100 with higher scores indicating better function. Changes in least squares mean (95% CI) from month 0 to month 4 are reported.
Time Frame: 4 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BA-LVR | ST-LVR
Number analyzed (Participants) | 87 | 76
units on a scale | 4.78 [1.34 to 8.21] | 2.36 [1.27 to 5.99]
Statistical Analysis 1: Comparison: BA-LVR vs ST-LVR; Test type: Superiority or Other; p = .34, Least squares mean; Mean Difference (Final Values) = 2.42, 95% CI 2-sided [-2.58 to 7.41]

5. Secondary Outcome: Quality of Life: Mental Health
Description: Self-reported menthal health was assessed using the Mental Health subscale from the National Eye Institute Vision Function Questionaire-25 (NEI-VFQ). Scores range from 0 to 100, with higher scores indicating better mental health. Changes in least square means from baseline to 4 months are presented.
Time Frame: 4 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BA-LVR | ST-LVR
Number analyzed (Participants) | 87 | 76
units on a scale | 2.23 [-3.2 to 7.66] | 4.25 [-1.32 to 9.81]
Statistical Analysis 1: Comparison: BA-LVR vs ST-LVR; Test type: Superiority or Other; p = .68, Least squares mean; Mean Difference (Final Values) = -2.02, 95% CI 2-sided [-9.80 to 5.76]

6. Secondary Outcome: Quality of Life: Role Functioning
Description: Self-reported role functioning was assessed using the Role Difficulties subscale from the National Eye Institute Vision Function Questionaire-25 (NEI-VFQ). Scores range from 0 to 100, with higher scores indicating fewer role difficulties . Changes in least square means from baseline to 4 months are presented.
Time Frame: 4 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BA-LVR | ST-LVR
Number analyzed (Participants) | 87 | 76
units on a scale | 2.33 [-1.46 to 6.12] | .93 [-2.96 to 4.82]
Statistical Analysis 1: Comparison: BA-LVR vs ST-LVR; Test type: Superiority or Other; p = .68, Least squares mean; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [-4.04 to 6.82]

7. Secondary Outcome: Quality of Life: Social Function
Description: Self-reported social function was assessed using the Social Functioning subscale from the National Eye Institute Vision Function Questionaire-25 (NEI-VFQ). Scores range from 0 to 100, with higher scores indicating better social function. Changes in least square means from baseline to 4 months are presented.
Time Frame: 4 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BA-LVR | ST-LVR
Number analyzed (Participants) | 87 | 76
units on a scale | -.38 [-5.59 to 3.84] | -2.00 [-7.46 to 3.47]
Statistical Analysis 1: Comparison: BA-LVR vs ST-LVR; Test type: Superiority or Other; p = .68, Least squares mean; Mean Difference (Final Values) = 1.62, 95% CI 2-sided [-5.94 to 9.17]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | BA-LVR | ST-LVR
Serious Adverse Events (participants affected / at risk) | 30/96 | 28/92
Other Adverse Events (participants affected / at risk) | 11/96 | 5/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BA-LVR (N=96) | ST-LVR (N=92)
death NOS (General disorders) | 5 (5) | 4 (4)
Stroke/TIA (Vascular disorders) | 8 (8) | 3 (3)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Cardiac (Cardiac disorders) | 2 (2) | 3 (3)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Break/fracture (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9)
GI (Gastrointestinal disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BA-LVR (N=96) | ST-LVR (N=92)
falls with no break/uti (General disorders) | 11 (11) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No